CLINICAL TRIAL: NCT03390036
Title: Trial Extension Protocol to Add a 39 Week Follow Up to Cingal 16-02, a Randomized, Double-Blind, Active Comparator Controlled, Multi-Center Study of a Single Injection of Cingal to Provide Symptomatic Relief of Knee Osteoarthritis
Brief Title: Study of Cingal for the Relief of Knee Osteoarthritis Compared to Triamcinolone Hexacetonide at 39 Weeks Follow up
Acronym: Cingal17-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cingal 17-02
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Intra-articular Injection; Hyaluronic Acid; Triamcinolone Hexacetonide
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — 3,6,9,16,19,22-hexaaza-6,19-bis(2-hydroxyethyl)tricyclo(22,2,2,2(11,14))triaconta-1,11,13,24,27,29-hexaene; triamcinolone hexacetonide

STUDY DESIGN:
Intervention Model Description: In the 16-02 study, subjects were randomized in a 4:4:1 ratio into the Cingal, Monovisc (hyaluronic acid) or TH (triamcinolone hexacetonide) arm. The 17-02 study is a 39-week follow-up to the 16-02 study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Study subjects and the Outcomes Assessor are blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cingal (Experimental): Cingal is a combination product consisting of 88 milligrams of crosslinked HA (hyaluronic acid) with 18 milligrams of TH (triamcinolone hexacetonide) in a 4 milliliter (mL) intra-articular injection.
  Interventions: Combination Product: Cingal
- Monovisc (Active Comparator): Monovisc is a device that consists of 88 milligrams of cross-linked HA (hyaluronic acid) in a 4 milliliter (mL) intra-articular injection.
  Interventions: Device: Monovisc
- Triamcinolone Hexacetonide (TH) (Active Comparator): Triamcinolone hexacetonide (TH) is a corticosteroid supplied in a 20 milligram per 1 milliliter (20 mg/mL) intra-articular injection.
  Interventions: Drug: Triamcinolone Hexacetonide

INTERVENTIONS:
Combination Product: Cingal — Hyaluronic Acid with Triamcinolone Hexacetonide
  Other Names: HA + TH
  Arms: Cingal
Device: Monovisc — Hyaluronic Acid
  Other Names: HA
  Arms: Monovisc
Drug: Triamcinolone Hexacetonide — Triamcinolone Hexacetonide
  Other Names: TH
  Arms: Triamcinolone Hexacetonide (TH)

SUMMARY:
Extension study to Cingal 16-02 to obtain 39-week safety and efficacy follow-up data

DETAILED DESCRIPTION:
Extension Study to Cingal 16-02: Trial Extension to 39 Week Follow Up in the Randomized, Double-Blind, Active Comparator Controlled, Multi-Center Study of a Single Injection Cross-Linked Sodium Hyaluronate Combined with Triamcinolone Hexacetonide (Cingal) to Provide Symptomatic Relief of Osteoarthritis of the Knee

ELIGIBILITY:
Inclusion Criteria:

1. Only subjects that were enrolled and met the inclusion criteria for the Cingal 16-02 trial and signed the informed consent are eligible for Cingal 17-02 trial.
2. Subject is able to understand and comply with the requirements of Cingal 17-02 and voluntarily provides consent.

Exclusion Criteria:

Patients will not be rescreened at enrollment to Cingal 17-02 as these patients met the inclusion / exclusion criteria for the Cingal 16-02 clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Hangody, MD, Principal Investigator — Uzsoki Hospital, Department of Traumatology
Locations (17):
- Hungary (7):
  - Health Center of Downtown-Lipotvaros, Orthopedic Outpatient Clinic (Belvárosi-Lipótvárosi Egészségügyi Szolgálat Ortopeadia), Budapest
  - Uzsoki Hospital, Department of Traumatology, Budapest
  - Jutrix Medical Llc, Budapest
  - Magyar Honvedseg, Egeszseugyi Kozpont, Balesteti Sebeszeti Osztaly, Budapest
  - DE KK Ortopediai Klinika, Debrecen
  - Medidea Bt., Kiskunfélegyháza
  - Kastelypark Klinka, Tata
- Poland (10):
  - Zdrowie Osteo-Medic, Bialystok
  - Szpital Świętego Łukasza S.A., Bielsko-Biala
  - NZOZ Medi SPATX, Gliwice
  - Centrum Medyczne 4M Plus, Krakow
  - Medical University of Lodz, Lodz
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - NOVAMED Jackowiak Krajewski Spółka Jawna, Torun
  - Centrum Medyczne Amed Warszawa Targówek, Warsaw
  - ETG Network, Warsaw, Warsaw
  - ETG Network, Warsaw

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled in Cingal 16-02 were given the option to enroll in Cingal 17-02 for a 39-week follow-up. 233 subjects in the Cingal arm (95%), 230 subjects in the Monovisc arm (93%), and 63 subjects in the Triamcinolone Hexacetonide arm (90%) elected to enroll in the extension study.
Pre-assignment Details: No enrolled participants were excluded.
Period: Overall Study
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Started (Safety Population and ITT Population) | 233 | 230 | 63
Completed | 231 | 230 | 63
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH) | Total
Number analyzed (Participants) | 233 | 230 | 63 | 526
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (8.8) | 57.7 (8.9) | 59.2 (8.4) | 57.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 152 | 44 | 361
  Male | 68 | 78 | 19 | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 233 | 230 | 63 | 526
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline WOMAC Pain in Index Knee [Mean (Standard Deviation); unit: millimeters (mm)] — Baseline knee pain is measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score, a validated visual analog scale (VAS) ranging from 0 mm = No Pain to 100 mm = Maximum Pain. Lower scores indicate less pain.
  millimeters (mm) | 63.5 (11.1) | 63.7 (11.4) | 64.6 (10.9) | 63.7 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: OMERACT-OARSI Responder Rate at 39 Weeks
Description: The post treatment Responder Rate at 39 weeks is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder. The criteria for response are (1) improvement in pain or physical function ≥50% and an absolute change ≥20 mm; or (2) improvement of ≥20% with an absolute change ≥10 mm in at least two of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome.
Time Frame: 39 weeks
Population: Intent to Treat population
Measure: Number; unit: Percentage of subjects
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Percentage of subjects | 91.2 | 92.4 | 93.2
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.8106, ANOVA

2. Secondary Outcome: Change From Baseline in WOMAC Pain Score at 39 Weeks
Description: The change from baseline in knee pain as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score at 39 weeks post treatment comparing the Cingal group to the Triamcinolone Hexacetonide group. The WOMAC Pain Score is a validated visual analog scale from 0 to 100 mm, where a higher score is equal to a higher pain level. A negative number for the difference from baseline indicates improvement in pain. A greater negative difference from baseline indicates a better outcome.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Millimeters (mm)
  Change from Baseline in WOMAC Pain 39 Weeks | -46.3 (20.2) | -47.2 (18.6) | -43.6 (21.4)
  Baseline WOMAC Pain in mm | 63.3 (11.0) | 63.3 (11.3) | 63.8 (11.3)
  39 Week WOMAC Pain in mm | 17.0 (19.3) | 16.0 (18.6) | 20.1 (21.1)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.3007, ANOVA

3. Secondary Outcome: Change From Baseline in WOMAC Physical Function Score at 39 Weeks
Description: This endpoint compares the change of the WOMAC Physical Function Score from baseline to Week 39 between the Cingal and Triamcinolone Hexacetonide arms. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Score is a validated visual analog scale from 0 to 100 mm, where a higher score is equal to a higher degree of functional limitation. A negative number for the change from baseline indicates improvement in physical function.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Millimeters (mm)
  Change from Baseline WOMAC Function 39 Weeks | -42.5 (22.4) | -43.5 (20.7) | -41.1 (22.5)
  Baseline WOMAC Function | 60.8 (15.2) | 60.8 (15.8) | 61.8 (15.7)
  39 Week WOMAC Function | 18.4 (19.8) | 17.3 (18.6) | 20.7 (21.3)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.6354, ANOVA

4. Secondary Outcome: Change From Baseline in WOMAC Stiffness Score at 39 Weeks
Description: The change from baseline in knee stiffness as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Score at 39 weeks post treatment comparing the Cingal group to the Triamcinolone Hexacetonide group. The WOMAC Stiffness Score is a validated visual analog scale from 0 to 100 mm, where a higher score is equal to a higher degree of stiffness. A negative number for the change from baseline indicates improvement in knee stiffness.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Millimeters (mm)
  Change from Baseline in WOMAC Stiffness 39 Weeks | -39.8 (24.4) | -42.0 (22.4) | -38.0 (24.9)
  Baseline WOMAC Stiffness in mm | 57.7 (19.3) | 59.2 (18.1) | 57.9 (17.6)
  39 Week WOMAC Stiffness in mm | 17.9 (20.0) | 17.2 (18.6) | 19.9 (21.9)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.5754, ANOVA

5. Secondary Outcome: Change From Baseline in Total WOMAC Score at 39 Weeks
Description: The change from baseline as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score at 39 weeks post treatment comparing the Cingal group to the Triamcinolone Hexacetonide group. The Total WOMAC Score is determined from the SUM of the scores from the WOMAC Pain Score, the WOMAC Stiffness Score, and the WOMAC Physical Function Score, resulting in a final range for Total Score from 0 mm to 240 mm. A higher Total WOMAC Score indicates a higher overall degree of pain, stiffness and functional limitations. A negative number for the change from baseline indicates improvement in the Total WOMAC Score.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Millimeters (mm)
  Change from Baseline in Total WOMAC 39 Weeks | -128.4 (63.1) | -132.6 (56.6) | -122.7 (62.2)
  Baseline Total WOMAC in mm | 181.8 (40.6) | 183.4 (39.4) | 183.5 (38.4)
  39 Week Total WOMAC in mm | 53.4 (58.1) | 50.8 (54.6) | 60.8 (62.5)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.4759, ANOVA

6. Secondary Outcome: Change From Baseline in Patient Global Assessment at 39 Weeks
Description: Comparison of the change of the Patient Global Assessment from baseline to 39 weeks between the Cingal and Triamcinolone Hexacetonide arms (ITT population). The Patient Global Assessment is done by the subject, and answers the question "Considering all the ways the osteoarthritis in your index knee bothers you, what is your assessment of how much your knee is bothering you today?" The Patient Global Assessment is scored on a 0 to 100 mm visual analog scale, where a higher number means the patient is bothered to a higher degree. A negative number for the change from baseline indicates a reduction (improvement) in the assessment.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Millimeters (mm)
  Change from Baseline in Patient Global 39 weeks | -38.6 (25.4) | -38.2 (22.8) | -36.7 (28.0)
  Baseline Patient Global in mm | 57.0 (18.9) | 56.0 (18.6) | 58.2 (20.3)
  39 Week Patient Global in mm | 18.4 (19.8) | 17.8 (19.4) | 21.5 (22.1)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.5596, ANOVA

7. Secondary Outcome: Change From Baseline in Evaluator Global Assessment at 39 Weeks
Description: Comparison of the change of the Evaluator Global Assessment from baseline to 39 weeks between the Cingal and Triamcinolone Hexacetonide arms (ITT population). The Evaluator Global Assessment is done by the Blinded Outcomes Assessor, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee bothers him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a 0 to 100 mm visual analog scale, where a higher number means the Evaluator assesses that the patient is bothered to a higher degree. A negative number for the change from baseline indicates a reduction (improvement) in the assessment.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Millimeters (mm)
  Change from Baseline in Evaluator Global 39 eeks | -37.1 (21.3) | -37.7 (19.9) | -39.1 (22.1)
  Baseline Evaluator Global in mm | 52.9 (17.2) | 52.3 (17.7) | 56.6 (18.1)
  39 Week Evaluator Global in mm | 15.8 (16.5) | 14.6 (16.5) | 17.4 (15.6)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.4551, ANOVA

8. Secondary Outcome: The Usage of Rescue Medication (Acetaminophen) at Week 39
Description: The usage of rescue medication (number of pills of acetominophen) at Week 39 weeks post treatment in the Cingal group compared to the Triamcinolone Hexacetonide group.
Time Frame: 39 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
Number analyzed (Participants) | 233 | 230 | 63
Number of pills | 7.9 (39.5) | 6.0 (18.7) | 6.9 (22.8)
Statistical Analysis 1: Comparison: Cingal vs Triamcinolone Hexacetonide (TH); Test type: Superiority; p = 0.7931, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the 26 Week visit (the last one in the Cingal 16-02 study) through the 39 Week visit in the Cingal 17-02 extension study.
Description: The adverse event descriptions used are consistent with the clinicaltrials.gov definitions.
Arm/Group | Cingal | Monovisc | Triamcinolone Hexacetonide (TH)
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/230 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/233 | 0/230 | 0/63
Other Adverse Events (participants affected / at risk) | 20/233 | 19/230 | 6/63
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=233) | Monovisc (N=230) | Triamcinolone Hexacetonide (TH) (N=63)
Headache (Nervous system disorders) | 7 (7) | 6 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) — Backache
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Cingal 17-02, an extension study of Cingal 16-02, did not include a placebo arm, and was an all-active trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03390036/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT03390036/SAP_001.pdf